CLINICAL TRIAL: NCT03968432
Title: The Feasibility, Acceptability, and Preliminary Effectiveness of Parent Targeted Interventions in Vaccination Pain Management of Infants: A Pilot Randomized Control Trial (RCT)
Brief Title: Parent Targeted Interventions in Vaccination Pain Management of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Shokoufeh Modanloo, PhD Candidate, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H-04-18-405
Record Dates: First submitted 2019-05-13; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Procedural Pain
Keywords: Childhood Vaccination,; Knowledge Translation,; Pain management,; Parents.
MeSH Terms: conditions — Pain, Procedural; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Sham Comparator): Be Sweet to Babies Videos and Pamphlet. Be Sweet to Babies vaccination pain management videos showing parents how to use breastfeeding, upright secure holding, and a small volume of the sweet solution during vaccination will be used.
  Interventions: Behavioral: Be Sweet to Babies Videos and Pamphlet
- Intervention (Active Comparator): Be Sweet to Babies Videos, pamphlet, and MIAS&Q. MIAS&Q includes five questions and statements based on MI approach which was developed by the researcher and was reviewed further by a panel of parent representatives and HCPs representatives and the research team consisting of the supervisor and two Ph.D. committee members. This MIAS&Q intervention consists of four scaled questions and two open-ended questions and presents brief informative and affirmative questions and statements. This aims to help the parents reflect on their own thoughts, and support them to advocate for the use of the recommended pain management strategies during their infant's vaccination.
  Interventions: Behavioral: MIAS&Q; Behavioral: Be Sweet to Babies Videos and Pamphlet

INTERVENTIONS:
Behavioral: MIAS&Q — There were two interventions compared in this study: 1) Be Sweet to Babies Videos and Pamphlet; and 2) Be Sweet to Babies Videos, pamphlet, and MIAS&Q. The Be Sweet to Babies vaccination pain management videos and pamphlet were provided to all participants as this information is publicly available, and demonstrates the effectiveness of the evidence-based recommended vaccination pain management strategies for infants. In addition, a pamphlet was used which was developed in partnership with CHEO and Ottawa Public Health as a knowledge translation tool. Those in the intervention arm were also given MIAS&Q included five questions and statements based on the MI approach consisted of four scaled questions and two open-ended questions, aimed to present brief informative and affirmative questions and statements to help the parents reflect on their own thoughts and support them to advocate for the use of the recommended pain management strategies during their infant's vaccination.
  Other Names: MI based affirmation statements and questions
  Arms: Intervention
Behavioral: Be Sweet to Babies Videos and Pamphlet — The Be Sweet to Babies vaccination pain management videos and pamphlet will be provided to all participants. Be Sweet to Babies vaccination pain management videos showing parents how to use breastfeeding, upright secure holding, and a small volume of sweet solution during vaccination, will be used. This pamphlet is a knowledge translation tool previously developed in partnership with the Children Hospital of Eastern Ontario (CHEO) and Ottawa Public Health and has been publicly available on the Ottawa Public Health Website since June 2013. The content presented about pain management for infants during vaccination is the same information as the video.

SUMMARY:
The overall aim of this study is to investigate the feasibility, acceptability, preliminary effectiveness and sustainability of parent-targeted interventions for pain management during vaccination of infants. To achieve the goal, a two-phase pilot randomized control trial is planned. Study one, currently in the data collection phase, aims i) to evaluate the feasibility and acceptability of data collection tools, participants' recruitment procedures and implementation process of parent-targeted interventions prior to infant vaccination at two, four, or six months. ii) to evaluate the preliminary effectiveness of parent-targeted interventions prior to infant vaccination in promoting the use of pain management strategies during vaccinations of infants at two, four, or six months. iii) to identify the parent's knowledge, use, intention and recommendation to use the recommended pain management strategies, and facilitators and barriers influencing the implementation of the parent-targeted interventions during vaccinations of infants at two, four, or six months. Methods. This study is a prospective multi-faceted two-armed pilot randomized control trial (RCT). a pilot randomized control trial. The participants are parents of infants, recruited before the infants receive their 2, 4, or 6- month vaccinations, who responded to the online invitation and consent to participate in this study. Parents living in Canada and prior to the infant receiving one of the three vaccinations were invited to participate through an online recruitment process. A sample of 50 parent/infant dyads in each group of control and intervention is estimated to be sufficient to achieve the study's goals. The outcome measurements are being done by five brief study questionnaires; Brief information of the study goals and the researchers' affiliation followed by a hyperlink to the survey were posted on different online platforms. Eligible parents of infants who respond to the study invitation are being randomly allocated to 1 of 2 groups (Intervention and control). There are two interventions in the study one being compared: 1) Be Sweet to Babies Videos and Pamphlet; and 2) Be Sweet to Babies Videos, pamphlet, and MIAS&Q. After the intervention, the impact of the vaccination pain management video and brochure followed by MIAS&Q questions are being evaluated by a brief online survey exploring the use of pain management (breastfeeding or sucrose and upright secure holding) during infants' vaccination in both groups. Following that, the opinion of parents about the understandability, applicability, feasibility, and acceptability of this study are evaluated. All data are being collected electronically using REDCap survey tool. SPSS version 23.0 (SPSS Inc, Chicago, Illinois) will be used to perform all descriptive and inferential statistical analyses. NVivo version 11.0 (Qualitative data analysis Software; QSR International Pty Ltd) will be used for content analysis and descriptive statistical analysis and thematic analysis will be used for the analysis of the qualitative data.

DETAILED DESCRIPTION:
Early childhood vaccination is the most important public health intervention to protect against life-threatening infectious diseases worldwide. However, vaccinations are painful and result in distress and anxiety for infants and, in many cases, their parents. If vaccination pain is not addressed, this pain can lead to subsequent non-adherence with vaccination schedules, fears of needles and avoidance of health care. Clinical practice guidelines and high-quality synthesized evidence shows that breastfeeding, sucrose, and upright secure holding effectively reduce pain during vaccination in infants. Despite the evidence, these strategies are not consistently used in practice highlighting an important gap in translating this knowledge into practice. Aims. The overall aim of this study is to investigate the feasibility, acceptability, preliminary effectiveness and sustainability of parent-targeted interventions for pain management during vaccination of infants. To achieve the goal, a two-phase pilot randomized control trial is planned. Study one, currently in the data collection phase, aims i) to evaluate the feasibility and acceptability of data collection tools, participants' recruitment procedures and implementation process of parent-targeted interventions prior to infant vaccination at two, four, or six months. ii) to evaluate the preliminary effectiveness of parent-targeted interventions prior to infant vaccination in promoting the use of pain management strategies during vaccinations of infants at two, four, or six months. iii) to identify the parent's knowledge, use, intention and recommendation to use the recommended pain management strategies, and facilitators and barriers influencing the implementation of the parent-targeted interventions during vaccinations of infants at two, four, or six months. Methods. This study is a prospective multi-faceted two-armed pilot randomized control trial (RCT). a pilot randomized control trial. The participants are parents of infants, recruited before the infants receive their 2, 4, or 6- month vaccinations, who responded to the online invitation and consent to participate in this study. Parents living in Canada and prior to the infant receiving one of the three vaccinations were invited to participate through an online recruitment process. Parents were eligible if they have an infant scheduled to receive their 2, 4, or 6-month routine vaccination as per the childhood immunization schedule of the province the parents are living in, and they read, speak and understand English sufficiently to understand the videos and complete the surveys. A sample of 50 parent/infant dyads in each group of control and intervention is estimated to be sufficient to achieve the study's goals. The outcome measurements are being done by five brief study questionnaires; Baseline demographic questionnaire, Baseline knowledge questionnaire, Knowledge utilization questionnaire, Acceptability, and feasibility questionnaire. All recruited parents of infants before their 2, 4, or 6-month vaccination were invited to take part in a baseline survey, aimed to assess current awareness, previous use and future intent to use one of the recommended pain care strategies (breastfeeding, sucrose/other sweet solutions and holding). Different methods were taken for online recruiting of the participants. Brief information of the study goals and the researchers' affiliation followed by a hyperlink to the survey were posted on different online platforms. When participants clicked on the survey link, they were directed to a REDCap (Research Electronic Data Capture) survey.

If the respondents are not eligible, a brief message containing a thank-you note and explanation about their in-eligibility to continue the study was sent to them. However, if they meet the listed screening criteria, they are directed to the next page which is the study's consent form. They are invited to read the forms and provide online informed consent to participate in this study. They are then being directed to the next page which is the demographic questionnaires. A hyperlink directs participants to a brief survey asking questions about previous awareness and intention to use specified recommended pain management strategies in their infants' future immunization episodes. In addition, they were asked to provide an email address to be contacted for the following steps of the study. Eligible parents of infants who respond to the study invitation are being randomly allocated to 1 of 2 groups (Intervention and control) in a 1:1 ratio before the infants' 2, 4, or 6-months vaccination. Participants were stratified according to the infant's age of receiving the vaccine (two, four, or six months). There are two interventions in the study one being compared: 1) Be Sweet to Babies Videos and Pamphlet; and 2) Be Sweet to Babies Videos, pamphlet, and MIAS&Q. The Be Sweet to Babies vaccination pain management videos and pamphlet are provided to all participants. Those in the intervention arm is also be given MIAS&Q. Be Sweet to Babies vaccination pain management videos showing parents how to use breastfeeding, upright secure holding, and a small volume of the sweet solution during vaccination, are used. In addition, the pamphlet is a knowledge translation tool developed in partnership with the Children Hospital of Eastern Ontario (CHEO) and Ottawa Public Health. MIAS&Q includes five questions and statements based on MI approach consists of four scaled questions and two open-ended questions, aimed to present brief informative and affirmative questions and statements. After the intervention, the impact of the vaccination pain management video and brochure followed by MIAS&Q questions are being evaluated by a brief online survey exploring the use of pain management (breastfeeding or sucrose and upright secure holding) during infants' vaccination in both groups. Following that, the opinion of parents about the understandability, applicability, feasibility, and acceptability of this study are evaluated. All data are being collected electronically using REDCap survey tool. SPSS version 23.0 (SPSS Inc, Chicago, Illinois) will be used to perform all descriptive and inferential statistical analyses. NVivo version 11.0 (Qualitative data analysis Software; QSR International Pty Ltd) will be used for content analysis and descriptive statistical analysis and thematic analysis will be used for the analysis of the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Parents of infants,
* Recruited before the infants receive their 2, 4, or 6-month vaccinations,
* Respond to the online invitation,
* Consent to participate in this study
* Parents living in Canada
* Read, speak and understand English sufficiently to understand the videos and complete the surveys.

Exclusion Criteria:

* Parents who cannot understand, read or communicate in English
* Do not plan to have their infant vaccinated

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome: Feasibility and acceptability of study procedure | after the study completion (4 months after the baseline survey)
  This outcome will be measured by the numbers of completed consent forms, number of completed surveys, and number of lost-to-fallow-up people.

SECONDARY OUTCOMES:
The secondary outcome: increase in use of pain management strategies | After the intervention (2 months after the baseline survey)
  This will be measured by the number/proportion of vaccination episodes where any of the recommended pain management strategies are used in comparison with baseline and it will be recorded by a self-report survey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Modanloo S, Dunn S, Stacey D, Harrison D. The feasibility, acceptability and preliminary efficacy of parent-targeted interventions in vaccination pain management of infants: a pilot randomized control trial (RCT). Pain Manag. 2021 May;11(3):287-301. doi: 10.2217/pmt-2020-0072. Epub 2021 Feb 17. PMID 33593096